CLINICAL TRIAL: NCT06560242
Title: Tracking Early Emergence of Sound Perception Impairments in FXS With Multimodal fNIRS/EEG- Infant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Elizabeth Smith, Assistant Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K23HD109375 Aim2; K23HD109375 (NIH)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Speech Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech Sounds (Experimental): Participants listen to speech sounds while the investigators measure electrical and hemodynamic changes in the brain.
  Interventions: Other: Speech discrimination

INTERVENTIONS:
Other: Speech discrimination — Two different speech sounds are played at the same sound intensity.

SUMMARY:
Individuals with Fragile X Syndrome show differences in how they understand and learn language from infancy. They frequently have lifelong delays in speech and language as well. In addition, they experience other auditory symptoms, including being very sensitive to certain sounds as well as being more sensitive than others to loud sounds. The underlying brain activity for sound perception and speech learning in Fragile X is not well understood, especially in the infant and toddler years. This study uses behavioral assessment of speech and language abilities, neuroimaging, and hearing tests to understand how speech and hearing are different in children with Fragile X Syndrome.

DETAILED DESCRIPTION:
Fragile X Syndrome (FXS) is the leading monogenic cause of intellectual disability and autism and is associated with extremely high risk for early delays in speech and language. While infancy is essential for speech and language development, neural mechanisms for language impairments have been studied entirely in older children and adults with FXS. Therefore, markers for speech and language impairments are unavailable in infants and toddlers with FXS to predict severity, test potential mechanisms, and track response to intervention. The investigators have identified a hallmark brain-based phenotype of hyperresponsiveness to sounds in adolescents and adults with FXS. This fundamental alteration in cortical responses to sound could influence early language delays, but this phenotype has not been explored in infants or toddlers with FXS.

Specifically, in this study the investigators will use simultaneous EEG/fNIRS during presentation of simple speech, stories, and nonspeech sounds to quantify and localize auditory hypersensitivity and neural differentiation in 30 infants and toddlers, including 15 with FXS and 15 controls. Infants will complete visits at different ages, with possible visits at 6 months, 12 months, 18 months, and 24 months, so that changes with development can be tracked over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of Fragile X Syndrome, Typical Development, or History of Premature Birth
* able to sit independently
* English is spoken at home

Exclusion Criteria:

* For all participants: no seizures in the past 6 months
* For typical development group and Fragile X group: not born prior to 32 weeks gestation

Ages: 6 Months to 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mullen Scales of Early Learning | at 12 month, 18 month, and 24 month visits
  change in Mullen Scales scores (age-corrected) from baseline on all subscales, including Expressive Language, Receptive Language, FIne Motor, Gross Motor, and Visual Reception. T-Scores from the Mullen Scales of Early Learning (MSEL) have a mean of 50 and a standard deviation of 10. Range=20-80. Higher scores indicate more advanced developmental skills.
Changes in oxygenated and deoxygenated hemoglobin concentration in response to sounds in language regions of the brain | at 12 month, 18 month, and 24 month visits
  Relative increase in oxygenated versus deoxygenated hemoglobin for no sounds, low intensity sounds, and medium intensity sounds. Measured via functional Near Infrared Spectroscopy with optodes placed over frontal, temporal, and parietal language regions.
Changes in amplitude of mismatch negativity response during sound discrimination | at 12 month, 18 month, and 24 month visits
  Electroencephalography is measured over the scalp while participant listens to speech sounds with infrequent "oddball" stimuli. Amplitude of the P100 for all stimuli as well as amplitude of the mismatch negativity response (frequent minus infrequent response) as well as change in these metrics over development are tracked in all groups.
Changes in hearing thresholds | at 12 month, 18 month, and 24 month visits
  Hearing thresholds in dB as assessed using Conditioned Play Audiometry (CPA) or Visual Reinforced Audiometry (VRA) dependent on child age and developmental ability.
Otoacoustic Emissions (OAEs) | at 12 month, 18 month, and 24 month visits
  Signals produced by excitation of hair cells in cochlea are measured for a range of frequencies.
Changes in tympanometric pressure profile in the inner ear | at 12 month, 18 month, and 24 month visits
  Wide Band Tympanometry is completed to measure variability in tympanometric pressure for left and right ears that may affect hearing profile.
Changes in LENA vocalizations and conversational turns | at 12 month, 18 month, and 24 month visits
  LENA is a voice recording system and proprietary program that records a child's home language environment. This recording is then digitally processed to model aspects of the child's own vocalizations and those of others'.

SECONDARY OUTCOMES:
Sensory profile 2 Auditory Processing subtest | at 6 month, 12 month, 18 month, and 24 month visits
  parent-report measure of child's behavioral responses to sounds in their environment
Sensory Profile 2 Attentional subtest | at 6 month, 12 month, 18 month, and 24 month visits
  parent-report measure of child's awareness of and responses to sensory cues in their environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified information will be shared as required for NIH grant supported studies.
Supporting Information: Study Protocol